CLINICAL TRIAL: NCT06970548
Title: Dexamethasone As Adjuvant for Pre - emptiveTransversusAbdominus Muscle Plane Block In Patient Undergoing Bariatric Surgery
Brief Title: Dexamethasone As Adjuvant for Pre - emptiveTransversusAbdominus Muscle Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nehal Samir Esmail, Lecturer of Anesthesia, intensive care and pain management Faculty of Medicine, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bariatric surgery
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2022-05

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Levobupivacaine; 21-benzyloxy-9alpha-fluoro-16alpha-methylpregna-1,4-dien-11beta,17alpha-diol-3,20-dione

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): About 20 patients received Ultrasound-guided (USG-TAP) block with 40 ml of 0.375% levobupivacaine plus 8ml dexamethasone. All participants then evaluated preoperatively by multidisciplinary team consist of internal medicine, nutritionist, psychotherapist, surgeon and anesthetist. And also they received standard general anesthesia technique with endotracheal intubation and muscle relaxant.The patients will be given 1-2 mg of midazolam intra venous as a premedication about 20 min before induction of general anesthesia. Standard monitoring included continuous electrocardiography (ECG), pulse oximetry, capnography and noninvasive blood pressure. General anesthesia will be induced with propofol 1.5-2 mg/kg and fentanyl 3 μg/kg. Tracheal intubation will be facilitated by administration of cis-atracurium 0.1 mg/kg. Anesthesia will be maintained with isoflurane 1MAC, cis-atracurium 2 μg/kg/min and fentanyl 1 μg/kg/h.
  Interventions: Drug: Levobupivacaine
- Group B: Control Group (Active Comparator): About 20 patients received only (USG-TAP) by 40 ml 0.375% levobupivacaine.All participants then evaluated preoperatively by multidisciplinary team consist of internal medicine, nutritionist, psychotherapist, surgeon and anesthetist. And also they received standard general anesthesia technique with endotracheal intubation and muscle relaxant. The patients will be given 1-2 mg of midazolam intra venous as a premedication about 20 min before induction of general anesthesia. Standard monitoring included continuous electrocardiography (ECG), pulse oximetry, capnography and noninvasive blood pressure. General anesthesia will be induced with propofol 1.5-2 mg/kg and fentanyl 3 μg/kg. Tracheal intubation will be facilitated by administration of cis-atracurium 0.1 mg/kg. Anesthesia will be maintained with isoflurane 1MAC, cis-atracurium 2 μg/kg/min and fentanyl 1 μg/kg/h.
  Interventions: Drug: Levobupivacaine

INTERVENTIONS:
Drug: Levobupivacaine — To evaluate efficacy of addition of dexamethasone to levopubivacaine in tranversusabdominis plane block (TAP) in postoperative pain management, postoperative analgesic consumption, and patient comfort after laparoscopic bariatric surgery.
  Other Names: Dexamethazone

SUMMARY:
Pain following bariatric surgery can be quite troublesome and prolongs recovery. Although laparoscopic bariatric surgery is minimally invasive and involves small incisions over the anterior abdominal wall, postoperative pain is frequent . Most morbidly obese patients also have obstructive sleep apnea and associated with cardiac co-morbidities. Prolonged postoperative pain in them may lead to delay in early ambulation and performing deep breathing exercises.

DETAILED DESCRIPTION:
Pain following bariatric surgery can be quite troublesome and prolongs recovery. Although laparoscopic bariatric surgery is minimally invasive and involves small incisions over the anterior abdominal wall, postoperative pain is frequent.

This this increases incidence of deep vein thrombosis and risk of pulmonary complications respectively. Because postoperative recovery is directly associated with the intensity and duration of pain, it is imperative to reduce the postoperative pain as early as possible. A substantial component of pain experienced by patients undergoing laparoscopic surgery is somatic pain arising from the port sites over the abdominal wall.

Many methods have been suggested for reducing the postoperative abdominal wall pain such as port site instillation of local anesthetics, patient-controlled analgesia (PCA), epidural catheterization, and use of non-steroidal anti-inflammatory drugs (NSAIDS). Opioid analgesics to counter immediate acute postoperative pain are known to cause postoperative nausea and vomiting (PONV).

The average reported incidence of PONV in immediate postoperative period in patients undergoing bariatric surgery is between 30 and 50% [5]. This contributes to increased costs, increased length of stay, increased perioperative morbidity, and prolonged overall recovery [6]. Systemically administered opioids also depress respiratory drive, level of consciousness, and supraglottic airway muscle tone resulting in hypoxia and hypercapnia.

The TransversusAbdominis Plane (TAP) block is a loco-regional analgesia technique that consists of infiltrating a local anesthetic solution between the plane of the transversus-abdominis muscle and the internal oblique muscle, laterally at the level of the triangle of Petit. The sensory nerves of the abdominal wall pass through this plane. This technique produces long-lasting analgesia, between 24-36 hours.

ELIGIBILITY:
Inclusion Criteria:

- 40 patients with American Society of Anesthesiologists (ASA) grade I to II, 20 to 65 years of age scheduled for Laparoscopic Sleeve Gastrectomy.

Exclusion Criteria:

* patient refusal.
* Chronic alcoholism
* Chronic opioid usage
* ASA Grade 4 or more
* Chronic kidney disease
* Chronic liver disease
* Chronic obstructive pulmonary disease.
* Known allergy to study medications.
* Pregnancy.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Relief | from 0 hours to 6 hours after the procedure
  Patient's pain score will be assessed using visual analogue scale (VAS); scored from 0-10 (where 0=no pain and 10=the worst pain imaginable) during the recovery room (T0) and at one, three, and six hours (T1, T3, and T6) in the postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed hamody Hassan, Principal Investigator — Anesthesiology, Intensive care, and Pain Management, Faculty of Medicine, Sohag University
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided